CLINICAL TRIAL: NCT01644422
Title: A Prospective Multicentric Open Label Randomized Bio-Interventional Phase I/II Pilot Study To Evaluate Safety & Efficacy Of Autologous Human Platelet Lysate For Treatment Of Androgenetic Alopecia In Patients Undergoing Hair Transplant
Brief Title: Study To Determine Safety & Efficacy Of Autologous Human Platelet Lysate in Androgenetic Alopecia After Hair Transplant
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kasiak Research Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRPL/HPL-AGA/11-12/001B
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Study arm A (Other): Subjects will receive hair follicles transplants that are dipped in HPL before transplant
  Interventions: Biological: Autologous Human Platelet Lysate
- Study arm B (Other): Subjects will receive hair follicles transplants that are dipped in HPL before transplant; followed by one HPL injection one week after transplant
  Interventions: Biological: Autologous Human Platelet Lysate
- Control arm C (Other): Subject will receive Standard hair follicle transplant
  Interventions: Other: Standard hair follicle transplant

INTERVENTIONS:
Biological: Autologous Human Platelet Lysate — Study arm A subjects will receive hair follicles transplants that are dipped in HPL before transplant
  Arms: Study arm A
Biological: Autologous Human Platelet Lysate — Study arm B subjects will receive hair follicles transplants that are dipped in HPL before transplant; followed by one HPL injection
  Arms: Study arm B
Other: Standard hair follicle transplant — Control arm subject will receive Standard hair follicle transplant
  Arms: Control arm C

SUMMARY:
This is a multicentre, open label, randomized, pilot study to evaluate safety and efficacy of Human Platelet Lysate (HPL) in subjects with Androgenetic Alopecia undergoing hair transplantation. The study is being conducted at 2 centers in India. The primary endpoints are Increase in Hair Follicle viability after transplant, Improvement in Caliber & Density of hair and Improvement in Photographic assessment from randomization to end of study. The secondary endpoints are Physicians and Patients self assessment score.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects, aged between 18 to 50 years (both inclusive) and in general good health
* Subjects willing to refrain from other AGA treatments during the entire study duration
* Subjects who are willing to give informed consent and adhere to the study protocol

Exclusion Criteria:

* Subjects aged <18 or > 50 years
* Subjects with dermatological disorder of scalp that might interfere with study evaluation
* Subjects on Anti-coagulant therapy
* Subjects with clinically significant medical or psychiatric disease as determined by the investigator.
* Subjects unwilling to or unable to comply with the study protocol.
* Subjects taking concomitant therapy that might interfere with the study results in investigators opinion or participating in another trial in the past 30 days.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-10 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Improvement in Calibre & Density of Hair as assessed by Folliscope | Day 0, Month 2, End of Study - Month 4

SECONDARY OUTCOMES:
Photographic assessment | Day 0, Month 1, Month 2, Month 3, End of Study - Month 4

OTHER OUTCOMES:
Physician's assessment score | End of Study - Month 4
Patient's self assessment score | End of Study - Month 4

CONTACTS AND LOCATIONS:
Overall Officials: Rajendarsingh Rajput, Dr., Principal Investigator — Dr. Rajesh Rajput Hair Restore; Sandeep Sattur, Dr., Principal Investigator — Hairrevive
Locations (1):
- Kasiak Research Pvt Ltd, Thane, Maharashtra, India